CLINICAL TRIAL: NCT05425095
Title: Comparative Effects of Buteyko Exercise and Corpse-Pose Technique on Physical Health and Quality of Life in Post-Cardiac Surgery Patients
Brief Title: Comparative Effects of Buteyko Exercise and Corpse-Pose Technique on Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0322
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Post-Cardiac Surgery Patients
Keywords: Cardiac surgery; Buteyko breathing technique; Corpse pose; Yoga; Quality of life; Physical Health; Short-form health survey SF-36

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko Breathing Technique (Experimental): Group A
  Interventions: Other: Buteyko Breathing Technique
- Corpse-Pose Technique (Experimental): Group B
  Interventions: Other: Corpse-Pose Technique

INTERVENTIONS:
Other: Buteyko Breathing Technique — Group A will be treated with Buteyko Breathing Technique. Patient in a relaxed sitting position will ask to take a gentle breath in (2 sec), breath out (3sec) followed by pinching the nose with hands to hold the breath. The therapist will count the no. of seconds the patient can comfortably hold the breath until feels the need to breathe in again. Followed by releasing the nose and continue breathing.
  Arms: Buteyko Breathing Technique
Other: Corpse-Pose Technique — Group B will be treated with Corpse-Pose Technique for 15-20 min.
  Arms: Corpse-Pose Technique

SUMMARY:
Open-heart surgeries such as coronary artery bypass grafting and valve replacements have been used to improve patient outcomes related to cardiac symptoms, prolongation of life, and health-related quality of life. Recovery from cardiac surgery is not entirely determined by physical attributes and medical treatment, but social and psychological factors may also influence the process of postoperative short and long-term recovery. The objective of this study is to find out the Comparative Effects of Buteyko Exercise and Corpse-Pose Technique on Physical Health and Quality of Life in Post-Cardiac Surgery Patients. This study will be a Randomized controlled trial and will be conducted in Faisalabad institute of cardiology after ethical approval. The study will be completed within the duration of 10 months after approval of synopsis. Nonprobability convenience sampling technique will be used. The sample size of 46 patients will be taken: 25 post-cardiac surgery patients in each group with a 10% attrition rate. There will be two groups in this study one will be given with the Buteyko breathing technique and other will be provided with corpse-pose technique. Treatment protocol for both techniques will be 4 weeks with 3 sets per day. A pre assessment at week 1 and a final assessment at week 4 will be made by using SF-36 questionnaire. Data will be analyzed on SPSS-25.

ELIGIBILITY:
Inclusion Criteria:

* Stable Post-Op Cardiac Surgery Patients (Post-3 months)
* Both genders.
* Age 40-70.

Exclusion Criteria:

* Patients on other medications. (Corticosteroids)
* Patients with underlying severe medical conditions

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Short Form-36 Health Survey Questionnaire (SF-36) | 4 Week
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes. this questionnaire has 36 scoring. 1 is minimum score and 36 is highest score.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Muriam Ghani, MSPT-CP, Principal Investigator — Riphah International University
Locations (1):
- Cardiac Rehabilitation Centre of Faisalabad institute of cardiology Hospital, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Management of Physical Health Conditions in Adults with Severe Mental Disorders. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK534487/ PMID 30507109
- [Background] Haraldstad K, Wahl A, Andenaes R, Andersen JR, Andersen MH, Beisland E, Borge CR, Engebretsen E, Eisemann M, Halvorsrud L, Hanssen TA, Haugstvedt A, Haugland T, Johansen VA, Larsen MH, Lovereide L, Loyland B, Kvarme LG, Moons P, Norekval TM, Ribu L, Rohde GE, Urstad KH, Helseth S; LIVSFORSK network. A systematic review of quality of life research in medicine and health sciences. Qual Life Res. 2019 Oct;28(10):2641-2650. doi: 10.1007/s11136-019-02214-9. Epub 2019 Jun 11. PMID 31187410
- [Background] Chen DM, Yu WC, Hung HF, Tsai JC, Wu HY, Chiou AF. The effects of Baduanjin exercise on fatigue and quality of life in patients with heart failure: A randomized controlled trial. Eur J Cardiovasc Nurs. 2018 Jun;17(5):456-466. doi: 10.1177/1474515117744770. Epub 2017 Nov 30. PMID 29189045
- [Background] Grand N, Bouchet JB, Zufferey P, Beraud AM, Awad S, Sandri F, Campisi S, Fuzellier JF, Molliex S, Vola M, Morel J. Quality of Life After Cardiac Operations Based on the Minimal Clinically Important Difference Concept. Ann Thorac Surg. 2018 Aug;106(2):548-554. doi: 10.1016/j.athoracsur.2018.02.050. Epub 2018 Mar 23. PMID 29580777
- [Background] Shah CH, Brown JD. Reliability and Validity of the Short-Form 12 Item Version 2 (SF-12v2) Health-Related Quality of Life Survey and Disutilities Associated with Relevant Conditions in the U.S. Older Adult Population. J Clin Med. 2020 Feb 29;9(3):661. doi: 10.3390/jcm9030661. PMID 32121371
- [Background] Guzelhan Y, Ugurlucan M, Oztas DM, Beyaz MO, Unal O, Bektas N, Conkbayir C, Alpagut U, Bozbuga N. Anxiety and health-related quality of life after cardiac surgery. Arch Med Sci Atheroscler Dis. 2020 Apr 8;5:e27-e35. doi: 10.5114/amsad.2020.94376. eCollection 2020. PMID 33585722